CLINICAL TRIAL: NCT05527145
Title: Treatment of Spinal Stenosis and Spolilolisthesis With Percutaneous Interspinous Spacers. A Phase III Trial
Brief Title: Spinal Stenosis and Listhesis Treated With Percutaneous Interspinous Spacer: a Non-surgical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Alessandro Napoli, Associate Professor of Radiology and Interventional Radiology, Department of Radiological, Pathological and Oncological Sciences, University of Roma La Sapienza
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: URomLS-0137/22
Record Dates: First submitted 2022-08-02; First posted 2022-09-02 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Lumbar Spine Degeneration; Lumbar Spine Instability; Lumbar Spondylolisthesis; Lumbar Spinal Stenosis
Keywords: spondylolisthesis; lumbar spine stenosis
MeSH Terms: conditions — Spondylolisthesis; Spinal Stenosis | interventions — Minimally Invasive Surgical Procedures

STUDY DESIGN:
Intervention Model Description: investigator-initiated, prospective, phase III, randomized, controlled clinical trial At the 6-month follow-up, there is a possibility of cross- over from group B to group A. After crossover to surgery, the after-treatment of these patients will be as in group A.
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- surgery (Active Comparator): Oper or minimally invasive surgery
  Interventions: Procedure: Minimally invasive surgery
- percutaneous (Active Comparator): percutaneous non-surgical insertion of interspinous device
  Interventions: Procedure: Percutaneous Spacer

INTERVENTIONS:
Procedure: Minimally invasive surgery — Surgery with decompression. Central decompression of the stenotic segment with undercutting of the lateral recesses.
  Arms: surgery
Procedure: Percutaneous Spacer — percutaneous image guided outpatient procedure that enables interspinous spacer insertion and fusion
  Arms: percutaneous

SUMMARY:
Symptomatic lumbar spinal stenosis is the most common indication for spinal surgery. However, more than one-third of the patients undergoing surgery for lumbar stenosis report dissatisfaction with the results. On the other hand, conservative treatment has shown positive results in some cases. This trial will compare the outcomes of surgical versus non-surgical treatment for lumbar stenosis.

DETAILED DESCRIPTION:
This is a three-centre randomised controlled trial in which 200 patients with symptomatic lumbar spinal stenosis will be randomised into one of two treatment arms. The patients in the surgical arm will undergo decompression of the neural structures by use of any open or minimally invasive (MIS) technique with or without fusion; the patients in the non-surgical arm will undergo imaging assisted percutaneous interspinous spacer insertion with fusion.

The primary outcome of the study will be the Oswestry Disability Index. Secondary outcomes will include motor amplitude and degree of denervation activity obtained by means of nerve conduction studies and electromyography.

Patient-reported outcome measures will be also used as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50-85 years.
2. Clinical symptoms of lumbar spinal stenosis (pseudoclaudication) indicating and motivating surgery. Numeric Rating Scale in lower limbs ≥3.
3. MRI with finding of lumbar spinal stenosis at 1-3 lumbar levels. Dural sac area ≤75 mm2 or degree of stenosis C or D according to Schizas's classification.34
4. The patient has given oral and written informed consent to participate.

Exclusion Criteria:

1. Degenerative deformity with Cobb angle >20°.
2. Symptomatic osteoarthritis in the lower limbs that affects and limits the patient's function.
3. Arterial insufficiency (claudication intermittent).
4. Former lumbar surgery other than disc hernia.
5. Conditions that affect the spine, such as ankylosing spondylitis, diffuse idiopathic skeletal hyperostosis, spondylodiscitis/infections, malignancy and neurological diseases.
6. Heart and lung diseases presenting a significant risk for surgery or making it impossible for the patient to take part in a percutaneous arm of treatment (American Society of Anesthesiologists (ASA) score >3).
7. Polyneuropathies.
8. Psychological factors rendering the patient incapable of inclusion in the trial (eg, drug addiction, dementia).

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
oswestry disability Index | 26 weeks
  system based on a % scale, with higher scores indicating greater disability; clinically important difference to improvement: 10%
oswestry disability Index | 52 weeks
  system based on a % scale, with higher scores indicating greater disability; clinically important difference to improvement: 10%

SECONDARY OUTCOMES:
Euro Quality of life Five-Dimensional descriptive system questionnaire (EQ-5D) | 26 and 52 weeks
Numeric Rating Scale (NRS) | 26 and 52 weeks
  for low back and leg pain (0-10 being 10 worst)
subjective walking ability tool | 26 and 52 weeks
neurophysiological measurements (NCSs/EMG) | 52 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Sapienza University of Rome, Policlinico Umberto I Hospital, Rome, Italy